CLINICAL TRIAL: NCT04601636
Title: Comparison of Continuous Active Prewarming Using Flex Warming Gown (3M) Versus Standard Care to Prevent Perioperative Hyporthermia in Short Outpatient Surgery Under General Anesthesia
Brief Title: Comparison of Active Prewarming Versus Standard Care to Prevent Perioperative Hyporthermia in Short Outpatient Surgery Under General Anesthesia
Acronym: PREWARMING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, Professor, MD, PhD, DESAR, Chair of Research, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-2427
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Hypothermia Following Anesthesia; Hypothermia, Accidental
Keywords: Outpatient Surgeries; Short Surgeries; Active Prewarming
MeSH Terms: conditions — Hypothermia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Prewarming group (PW group) (Active Comparator): Group randomized to receive at least 30 minutes of active prewarming before induction of anesthesia, combined to active warming intraoperatively.
  Interventions: Device: Active Prewarming
- Control group (C group) (Placebo Comparator): Group randomized to receive the standard care : passive prewarming before induction of anesthesia combined to active warming intraoperatively.
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: Active Prewarming — Active prewarming with Flex Warming Gown (Bair Paws, 3M) for at least 30 minutes before induction of anesthesia, with active warming intraoperatively with Bair Hugger (3M)
  Arms: Active Prewarming group (PW group)
Other: Standard Care — Standard care with a passive prewarming (warm cotton blankets) before induction of anesthesia, with active warming intraoperatively with (Bair Hugger, 3M)
  Arms: Control group (C group)

SUMMARY:
The purpose of this prospective randomized controlled study is to compare the efficiency in preventing perioperative hypothermia of a continuous active prewarming combined with active intraoperative warming versus passive prewarming plus intraoperative warming for short outpatient surgery.

DETAILED DESCRIPTION:
The prevalence of accidental perioperative hypothermia is high, ranging from 20 to 90% in the literature, and its prevention still remains a major issue despite the many existing prevention techniques. Perioperative hypothermia is defined as a core body temperature below 36.0 ° Celsius.

The deleterious effects of perioperative hypothermia are well known : increased risk of wound infection, adverse cardiac events and blood loss. Moreover, the pharmacology of anesthetic agents can be altered by hypothermia, which in turn could lengthen the emergence of anesthesia. Patient comfort and satisfaction are also related to hypothermia and the feeling of cold generated.

Thus, hypothermia may be associated with prolonged length of stay in the recovery room and in the hospital for outpatient surgeries. Therefore, hypothermia can indirectly increase the costs of an intervention.

Several techniques have been described for the prevention of perioperative hypothermia. Passive warming is a method used to prevent heat loss such as warm cotton blankets, drapes or plastics whereas active warming consist in adding heat to the body surface using a warming system such as forced-air warming to increase mean body temperature. So, the use of a prewarming, an active warming before induction of anesthesia, could reduce the potential for redistribution, the main mechanism of hypothermia under general anesthesia.

Based on a literature review, the combined use of active prewarming with intraoperative active warming appears to be the most effective technique in preventing hypothermia upon arrival in the recovery room for inpatient surgeries lasting longer than 30 minutes. In the literature, the majority of publications on prewarming focus on surgeries lasting at least one hour, despite strong recommendations to use active warming for surgeries of 30 minutes or more. There is not so much data regarding the efficiency of continuous prewarming for short outpatient surgeries, from the preoperative unit to induction of anesthesia.

This prospective randomized controlled study is designed to evaluate if the combination of a continuous active prewarming of at least 30 minutes (Flex Warming Gown, Bair Paws, 3M) with an active intraoperative warming (Bair Hugger, 3M) would be effective in demonstrating a significant difference in temperature at the end of surgery between the two groups (control and intervention) for short (30 to 120 minutes) outpatient surgeries under general anesthesia. This intervention will be compared to the standard care which are a passive warming preoperatively with an active intraoperative warming.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status I to III
* Elective Outpatient Surgery under General Anesthesia
* Surgery Length from 30 to 120 minutes (from induction of anesthesia to extubation)

Exclusion Criteria:

* Patient refusal or inability to consent
* Neuraxial (spinal or epidural) anesthesia
* BMI over 40 (Flex gown limitation)
* Pregnancy
* Active infection
* Systemic disease which impairs thermoregulation (hypothyroidism or hyperthyroidism, adrenal insufficiency, major burns, para / quadriplegia)
* Medications affecting core body temperature (like levothyroxine)
* Facial surgery
* Use of a fluid warmer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Temperature at the end of surgery (°Celsius) | Measure taken at the end of surgery, before the patient leaves the operating room for the recovery room (below 120 minutes)
  Patient Temperature at the end of surgery

SECONDARY OUTCOMES:
Incidence of Hypothermia (presence or absence) | Intraoperative (time frame when patient is in the operative room - below 120 minutes)
  Incidence of hypothermia, defined as a core body temperature below 36°Celsius
Delta Temperature Loss (°Celsius) | Intraoperative (time frame when patient is in the operative room - below 120 minutes)
  Maximum Temperature Loss intraoperatively (from the temperature at entry in the operating room to the minimum temperature reached during surgery )
Shivering incidence (number of episodes) | Length of Stay in the Recovery Room (maximum 2h)
  Number of shivering episodes at the recovery room
Grade of Shivering (likert scale 0 to 4) | Length of Stay in the Recovery Room (maximum 2h)
  Grade of Shivering according to Crossley and Mahajan grading scale of intraoperative shivering (from 0 to 4)
Recovery Room Length of Stay (minutes) | Length of Stay in the Recovery Room (maximum 2h)
  Length of Stay in the Recovery Room
Patient Comfort Level (likert scale 0 to 10) | Right before entry in the operating room
  Evaluation of the Patient's Thermal Comfort Level according to a verbal numerical rating scale (from 0 - extremely uncomfortable ; to 10 - extremely comfortable)

CONTACTS AND LOCATIONS:
Locations (1):
- CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada